CLINICAL TRIAL: NCT06343818
Title: The Compassion Project: Developing and Piloting an Intervention to Reduce Empathy-Based Stress on Adolescent Mental Health Wards
Brief Title: Compassion Project: Developing an Empathy-Based Stress Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Oxford Health NHS Foundation Trust (Other Government); Central and North West London NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Lucy Maddox, Principal Investigator, University of Bath
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NIHR301578
Record Dates: First submitted 2024-03-15; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Reduction of Empathy-Based Stress in Healthcare Staff
Keywords: Compassion Fatigue; Burnout; Secondary Trauma; Empathy-Based Stress; Staff wellbeing; Patient care
MeSH Terms: conditions — Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The study uses a repeated AB design on two ward sites to assess feasibility, acceptability and usefulness of a novel intervention for empathy-based stress in staff, and to test feasibility of this study design. It is not assessing efficacy. The extended baseline measure is the control, there is no control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Ward Site 1 (Experimental): First ward site will pilot the intervention which will then be refined before delivery at second ward site
  Interventions: Other: The Compassion Project: Intervention to Reduce Empathy-Based Stress in Staff
- Pilot Ward Site 2 (Experimental): Second ward will pilot refined intervention
  Interventions: Other: The Compassion Project: Intervention to Reduce Empathy-Based Stress in Staff

INTERVENTIONS:
Other: The Compassion Project: Intervention to Reduce Empathy-Based Stress in Staff — Six month package of training and resources delivered to ward staff, including bite-sized audio, video and written materials. Face to face training will be provided weekly by a clinical psychologist. A staff group of 'compassion champions' will be responsible for embedding the intervention.

SUMMARY:
Compassion is recognising that someone is suffering and wanting to help them. Compassion fatigue is a reduction in capacity to feel compassion for others. Secondary trauma is the experience of traumatic responses to hearing about someone else's trauma. Burnout is depersonalisation, emotional exhaustion, and feeling less good at one's job. Compassion fatigue, secondary trauma and burnout can all be referred to as empathy-based stress. This is a problem for healthcare staff and their patients.

Staff experiencing empathy-based stress deliver less high quality care, which can lead to serious consequences for patients. Empathy-based stress is also associated with staff sickness, which is bad for staff and costly to the United Kingdom's National Health Service (NHS).

Child and adolescent mental health (CAMHS) wards are busy, high-pressure environments where families and young people are often upset, resources are stretched, and staff are managing high levels of patient risk of self-harm or suicide.

The principal investigator has already reviewed research on empathy-based stress and interventions to prevent and/or reduce it in mental health ward staff. This evidence has been presented to CAMHS ward staff, managers, commissioners, patients and families and these stakeholders have co-designed an intervention for wards, to reduce empathy-based stress. The intervention aims to help staff to feel better and care better.

This pilot study aims to test and improve our intervention on two CAMHS wards, measuring how useful and well-liked it is, and how feasible it would be to use it and to test it on more wards. Staff on CAMHS wards will be offered a modular intervention including psychoeducation about empathy based stress and ways of combatting it, and workplace stressor and management toolkits. NHS CAMHS ward staff and patients will be asked to complete questionnaires and a subsample of staff will be asked to complete interviews about the process of the intervention.

DETAILED DESCRIPTION:
A novel intervention aiming to reduce empathy-based stress in staff will be piloted sequentially on two adolescent mental health wards. After delivery on the first ward, feedback from post-intervention questionnaires and interviews with a subsample of staff will be used to modify the intervention before delivery on the second ward. The study aims to assess acceptability, usefulness and feasibility of the intervention, and feasibility of using these study methods (with a view to potentially trialing this intervention at a later date).

The intervention is called The Compassion Project, and it is a 6 month package which aims to target individual staff understanding and coping responses and also organisational practices. The Compassion Project uses a multi-level approach incorporating staff training, a range of resources and support for staff. These will include training materials (in audio, video and written forms), opportunities to discuss how current ward practices could be improved and to celebrate those which are working well. This intervention involves a modular structure encompassing individual, team and more organisational (through targeting management staff) levels of intervention. A working group of Compassion Champions from all levels of ward staff groups will work to embed the principles in the ward's practice. The intervention has been developed using information from a systematic literature review, Intervention Mapping and co-design with stakeholders.

The study uses a repeated AB design. Repeated baseline (A) and post-intervention (B) measures will be collected, then this will be repeated on the second ward. A mid-point measure will also be collected. The four measurement timepoints are -1 month, 0 months, 3 months and 6 months for staff to complete questionnaires. In addition, young people and parents/carers cared for by the ward at the time of intervention will be asked to complete two questionnaires at the point of discharge. Ward level measures (e.g. number of incidents) will allow context to be understood and also capture any changes over the course of the intervention, they will contribute to economic analyses also.

ELIGIBILITY:
Inclusion Criteria:

* Staff working on the 2 adolescent mental health ward sites at this time. All young people and parents/carers who are discharged during the time period of the intervention.

Exclusion Criteria:

* There are no exclusion criteria for staff. For young people who are inpatients on the ward and parents/carers of young people, an exclusion criteria would be if levels of English are such that questionnaires are inaccessible without reasonable adjustments and a supporting person is not available. We will strive to include all potential participants in the study if supporters are available to help an individual access the questionnaires.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention | Month 3 and Month 6
  Acceptability of Intervention Measure (AIM), with a minimum score of 1 and a maximum score of 15, with higher scores indicating greater acceptability.
Feasibility of intervention | Month 3 and Month 6
  Feasibility of Intervention Measure (FIM), with a minimum score of 1 and a maximum score of 20, with higher scores indicating greater perceived feasibility.
Perceived usefulness of intervention | Month 3 and Month 6
  Two perceived usefulness questions rated on a 5 point Likert scale where 1 is not useful and 5 is extremely useful
Feasibility of Study | Conducted in month 6
  Red/Amber/Green analysis of ward recruitment
Feasibility of gathering data on staff empathy-based stress using the Professional Quality of Life Scale at multiple timepoints | Month -1, 0, 3 and 6
  Professional Quality of Life Scale (PROQUOL). Raw scores between 10 and 50 are presented for three subscales (1) Compassion Satisfaction, (2) Burnout and (3) Secondary Traumatic Stress. Higher scores on compassion satisfaction are positive, and higher scores on burnout or secondary traumatic stress relate to a poorer outcome.

SECONDARY OUTCOMES:
Feasibility of assessing health economics data using a Health-related Quality of Life questionnaire | Month -1, 0, 3 and 6
  European Quality of Life 5 Dimensions 5 Level Version (EQ5D-5L) Questionnaire
Process measures to assess potential mechanisms of change | Month -1, 0, 3 and 6
  Knowledge about empathy-based stress questionnaire devised for the study (greater scores indicate greater knowledge) Mindful Attention and Awareness Scale (MAAS) (mean scores range from 1-6, with greater scores indicating greater mindfulness) Self-Compassion Scale (SCS) (minimum score is 1, maximum score is 60, with higher scores indicating more self compassion) Health and Safety Executive (HSE) Management Standards Questionnaire Questions about training Subsample of 15 qualitative interviews about process of the intervention
Feasibility of gathering young person and parent/carer data on compassionate care | Given at discharge throughout the 6 months of the intervention
  A questionnaires relating to care will be administered to young people and parents/carers on discharge. This is the Sinclair compassion Questionnaire Short Form
Feasibility of gathering young person and parent/carer data on experience of service | Given at discharge throughout the 6 months of the intervention
  Two questionnaires relating to care will be administered to young people and parents/carers on discharge. This is the Experience of Service Questionnaire.

OTHER OUTCOMES:
Ward-level contextual factors | Month -1, 0, 3 and 6
  Ward level contextual factors (e.g. number of incidents) will allow context to be understood and also capture any changes over the course of the intervention. Ward data will be gathered on ward caseload (ward occupancy), length of stay of patients, incidents on the ward, staff sickness, number of staff leaving. These will be collected using a data sheet filled in by ward modern matrons using readily available data

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Maddox, DClinPsy, Principal Investigator — University of Bath

IPD SHARING:
Plan to Share IPD: No
Amalgamated data will be stored in a data repository and made available to researchers if they have a good reason to request it. All data will be anonymised and individual data will not be recognisable.